CLINICAL TRIAL: NCT02188849
Title: Effects of Creatine Supplementation on Muscle Mass and Function Among Older Women Subjected to Resistance Training
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Daniel Bunout, Medical Doctor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Creatine elderly; Creatine INTA (Other: INTA U de Chile)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Muscle Weakness
Keywords: creatine; resistance training; older women; muscle strength
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training; Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Creatine (Experimental): Creatine 5 g/ day
  Interventions: Other: Resistance exercise training; Drug: Creatine
- Placebo (Placebo Comparator): Maltodextrin 5 g/day to be dissolved in water
  Interventions: Other: Resistance exercise training

INTERVENTIONS:
Other: Resistance exercise training — All participants will be subjected to resistance training of upper and lower limbs, using elastic bands and tubing and free weights. Training will be calibrated at 60% of one repetition maximum for each muscle group with three sets of 15 repetitions with one minute rest between each set. All exercises will be additionally calibrated to be of moderate intensity according to the Borg scale. The exercise load will be adapted according to the progression of each participant.
Drug: Creatine — Creatine powder 5 g day
  Arms: Creatine

SUMMARY:
To determine, in a double blind trial, the effects of creatine supplementation during 12 weeks on muscle mass and function of community living older women subjected to resistance training. Material and methods: Fifty healthy older women will be selected for the study. All participants will be subjected to a progressive resistance training program using elastic bands and weights, consisting in three sessions per week lasting 1 hour. Participant will be randomly allocated in a double blind fashion, to receive creatine 5 g per day or an identical placebo. The training and supplementation period will last 12 weeks. At baseline and at the end of the study, body composition will be measured by dual energy x-ray absorptiometry, rectus femoris cross sectional height and surface will be measured by ultrasound, quadriceps strength will be measured in a quadriceps table and 12 minutes' walk will be assessed. The main outcome measure will be quadriceps cross sectional height. Expected results: We expect that creatine supplementation will increase rectus femoris height over and above the effect of resistance training.

DETAILED DESCRIPTION:
Healthy women of middle and low socioeconomic level, living in the community and aged between 60 and 75 years, will be invited to participate in this study.

At baseline and after signing an informed consent form, the following assessments will be carried out:

1. A complete medical history including medications, previous diseases and surgical procedures.
2. Evaluation of usual physical activity using the International Physical Activity Questionnaire (IPAQ) .
3. Minimental state examination .
4. Mininutritional assessment .
5. Measurement of weight, height, waist and hip circumference.
6. Measurement of body composition by double energy X ray absorptiometry in a General Electric iDEXA equipment.
7. Measurement of rectus femoris cross sectional height using a General Electric LogiQ ultrasonographer. Measurements will be made with the participant in supine position and the tight relaxed. The mid-point between the superior anterior iliac spine and the superior border to the patella will be the measurement point.
8. Measurement of quadriceps isometric force using a quadriceps table as previously described .
9. Measurement of hand grip strength using a hand grip dynamometer.
10. Measurement of 12 minutes walking capacity .

After performing the baseline assessment, participants will be randomized in one of two groups, balancing by age and nutritional status, using a double blind design:

1. The active group will receive creatine 5 g/day in one dose as a powder to be dissolved in water
2. The control group will receive a placebo of similar aspect and taste as creatine.

The active prescription and the placebo will be identified by a unique numeric code. The codes will be known by an external professional, not involved in the research. In case of adverse events, the opening of a specific patient code of a will be requested to this professional, who will decide the pertinence of the request. Thus, even breaking one code, the double blind will be maintained for the rest of participants

All participants will be incorporated to an exercise training program, that will last 12 weeks, with three sessions per week. Each exercise session will consist of:

1. A warm-up period of 15 minutes, consisting in walking and cycling in braked bicycle ergometers.
2. Resistance training of upper and lower limbs, using elastic bands and tubing and free weights. Training will be calibrated at 60% of one repetition maximum for each muscle group with three sets of 15 repetitions with one minute rest between each set. All exercises will be additionally calibrated to be of moderate intensity according to the Borg scale. The exercise load will be adapted according to the progression of each participant.
3. An elongation period lasting 10 minutes that will include elongation in mats and exercise balls.

The attendance of participants to each session, their level of engagement with the exercise protocol and the overall Borg score will be recorded. All adverse events will be also recorded following good clinical practice guidelines Every two weeks, a new supply of the research prescription will be delivered. Participants will be requested to return the unused sachets to have an approximate assessment of compliance.

At the end of 12 weeks of intervention, all the assessments done at baseline will be repeated.

All the information of participants will be recorded in encrypted INTERNET databases. Only researchers will have access to the information, but participants will be informed about the results of all assessments.

Main outcome measure and calculation of sample size:

The main outcome will be rectus femoris cross sectional height. According to previously published results, this parameter increases from 20 ± 3.2 to 24.3 ± 3.8 mm after a training period of 12 weeks . If we expect a 15% difference in rectus femoris cross sectional height at the end of the intervention period, we would require 19 participants per group to obtain differences with an α of 0.05 and a power of 0.8- Considering an attrition rate of 30% during training, we would require 25 participants per group.

Analysis of results:

An intention to treat analysis will be performed. Also a safety analysis will also be carried out, considering all participants that took at least one dose of creatine or placebo. According to the normality of variable distribution, parametric or non-parametric tests will be used to analyze differences.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of a significant disability, defined as the capacity to reach the health center by their own means with the use of any aid such as canes or wheelchairs
2. Absence of disabling diseases such as cardiac, respiratory, liver or kidney failure or active cancer
3. Absence of decompensated diabetes mellitus of hypertension. Diabetic patients with repeated fasting blood glucose levels below 120 mg/dl and a glycosylated hemoglobin below 7% will be allowed to participate. Hypertensive patients in treatment with a blood pressure (measured in at least two occasions) below 140/90 mm Hg will also be allowed.

Exclusion Criteria:

1. Smoking or excessive consumption of alcohol
2. Use of medications that can cause muscle dysfunction or limit exercise capacity such as adrenal steroids, chemotherapeutic agents, statins in high doses (ie more than 40 mg/day of atorvastatin) or muscle relaxants.
3. Having a severe osteoarticular disease such as rheumatoid arthritis or severe osteoarthritis, with precludes participating in an exercise training program.
4. Recent use of ergogenic supplements such as creatine.
5. Being engaged in an active exercise training program.
6. Being illiterate or having a level of cognitive dysfunction that precludes the free signature of a written informed consent to participate in the study.
7. Any personal or socioeconomic condition that, in opinion of the research team, will hamper the correct compliance of the participant with the research program.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Hirsch, MD, Study Director — INTA University of Chile
Locations (1):
- INTA University of Chile, Santiago, Metropolitan, Chile

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Creatine | Placebo
Started | 25 | 25
Completed | 22 | 17
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Creatine | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (4.5) | 68.1 (4.9) | 67.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Chile | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Rectus Femoris Cross Sectional Height
Description: Measurement of rectus femoris cross sectional height in the mid thigh by ultrasound
Time Frame: Twelve weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Creatine | Placebo
Number analyzed (Participants) | 22 | 17
cm | 17.5 (2.0) | 17.6 (2.8)

2. Secondary Outcome: Quadriceps Isometric Strength
Description: Measurement of quadriceps isometric force using a quadriceps table
Time Frame: Twelve weeks
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Creatine | Placebo
Number analyzed (Participants) | 22 | 17
Newtons | 278.6 (53.9) | 225.3 (50.6)

3. Secondary Outcome: Twelve Minutes Walk
Description: Measurement of the distance that a participant can walk during 12 minutes
Time Frame: Twelve weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Creatine | Placebo
Number analyzed (Participants) | 22 | 17
meters | 1091.4 (101.1) | 1087.5 (108)

4. Other Pre Specified Outcome: Serum Creatinine
Description: Serum creatinine levels
Time Frame: Twelve weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Creatine | Placebo
Number analyzed (Participants) | 22 | 17
mg/dl | 0.8 (0.12) | 0.75 (0.13)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Creatine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 11/22 | 8/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine (N=22) | Placebo (N=17)
Falls (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Gastroinftestinal symptoms (Gastrointestinal disorders) | 3 (4) | 2 (3)
Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6)
Fever (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No